CLINICAL TRIAL: NCT05812742
Title: Neurofilament Light Chain, Inflammatory Markers, Calcitonin Gene-related Peptide, and Kynurenine Metabolites in Patients With Severe Post-concussive Symptoms
Brief Title: Chasing Biomarkers in Post-concussion Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Sygekassernes Helsefond (Other); Fonden til Lægevidenskabens Fremme (Other); Direktør Emil C. Hertz og Hustru Inger Hertz Fond (Unknown); Helga Og Peter Kornings Fond (Unknown); Region MidtJylland Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Biomarkers in GAIN 1.0
Record Dates: First submitted 2023-03-01; First posted 2023-04-14 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2023-02

CONDITIONS: Post Concussive Symptoms
MeSH Terms: conditions — Post-Concussion Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care (Active Comparator): For more details on the intervention, please go to the original registration of the RCT-study (NCT02337101) or the published article (PMID: 31891145).
  Enhanced Usual Care (EUC) All patients had a brief clinical psychiatric and neurological assessment in order to determine eligibility, and they were provided with information and advice about typical post-concussional symptoms, the typical recovery process and the use of pain medication.
  Interventions: Behavioral: Enhanced usual care
- Enhanced Usual Care + Early intervention programme (Experimental): For more details on the intervention, please go to the original registration of the RCT-study (NCT02337101) or the published article (PMID: 31891145).
  Behavioral: EUC + Early intervention programme All patients had a brief clinical psychiatric and neurological assessment in order to determine eligibility, and were provided with information and advice about typical post-concussional symptoms, the typical recovery process and the use of pain medication.
  The early intervention programme was interdisciplinary and was provided by an occupational therapist and a physiotherapist under supervision of a neuropsychologist. It was based on psychoeducation and principles from Cognitive Behavioral Therapy and Graded Exercise Therapy and targeted to patients' individual goals.
  Patients received 8 weekly treatment sessions (3 group based and 5 individual sessions). The intervention started approximately 4 months after the concussion.
  Interventions: Behavioral: Early intervention programme; Behavioral: Enhanced usual care

INTERVENTIONS:
Behavioral: Early intervention programme — For more information, please go to the original registration of the RCT-study (NCT02337101) or the published article (PMID: 31891145).
  Arms: Enhanced Usual Care + Early intervention programme
Behavioral: Enhanced usual care — For more information, please go to the original registration of the RCT-study (NCT02337101) or the published article (PMID: 31891145).

SUMMARY:
The goal of this study was to investigate the biomarkers, neurofilament light chain, inflammatory markers, calcitonin-gene-related peptide, and metabolites from the kynurenine pathway in patients with severe post-concussive symptoms. The main question it aimed to answer was:

* Are the biomarker concentrations significantly changed in patients with severe post-concussive symptoms compared to healthy individuals?
* Do the biomarker concentrations change at follow-up?

Participants were recruited from a recently published randomized controlled trial (Clinicaltrials.gov no. NCT02337101 / PMID: 31891145 ). The biomarker concentrations were compared to a healthy control group recruited from the Blood Bank at Aarhus University Hospital in 2022.

DETAILED DESCRIPTION:
In the previously published RCT-study (PMID: 31891145), 86 participants with severe post-concussive symptoms provided blood samples at baseline (4 months after the concussion). Severe post-concussive symptoms were defined as having a Rivermead Post Concussion Questionnaire >20.

Around 7 months later, a follow-up blood sample was obtained from 54 participants.

These blood samples were used to investigate blood biomarkers for the condition.

ELIGIBILITY:
Patients with severe post-concussive symptoms:

Inclusion Criteria:

1. Concussion caused by a head trauma based on the diagnostic criteria recommended by the World Health Organization (WHO) Task Force
2. Age between 18 and 30 years
3. Able to understand, speak and read Danish.
4. A score of 20 or more on the Rivermead Post Concussion Symptoms Questionnaire (RPQ).

Exclusion Criteria:

1. Objective neurological findings indicating neurological disease or brain damage.
2. Previous concussion leading to persistent post-concussional symptoms within the last two years.
3. Severe misuse of alcohol, prescription drugs and / or illegal drugs.
4. Severe psychiatric, neurological,or other medical disease that would impede participation in the intervention
5. Inability to speak and read Danish

Healthy control group (recruited from December 2021 - March 2022):

- Individuals from the Blood Bank at Aarhus University Hospital in Denmark.

Inclusion criteria were:

1. Age between 18-30 years
2. Equal distribution between the genders (60 men and 60 women). This number was based on a power analysis using published data from neurofilament light chain.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2023-07 (Actual); Study Completion 2023-07 (Actual)

PRIMARY OUTCOMES:
Neurofilament light chain at baseline (primary outcome) | The baseline blood sample was taken up to 7 months after the concussion (4 months median).
  The investigators hypothesized:
  The concentration of neurofilament light chain (ng/L) is significantly increased at baseline in patients compared to the healthy control group.
Neurofilament light chain at follow-up (primary outcome) | The follow-up blood sample was taken up to 12 months after baseline (7 months median) after the baseline blood sample.
  The investigators hypothesized:
  1)The neurofilament light chain concentration (ng/L) normalizes (decreases) at follow-up compared to the baseline concentration in patients.
Self-reported post-concussion symptoms score (primary outcome) | The baseline symptom score (RPQ) was obtained from the patients up to 7 months after the concussion (4 months median), and the follow-up score was obtained up to 16 months (10.5 median) after the concussion
  The symptom score was measured at both baseline and follow-up using the Rivermead Post-Concussion Symptoms Questionnaire (RPQ) which is a self-reported questionnaire. The Rivermead Post-Concussion Symptoms Questionnaire contains 16 items which is rated from 0 (not experienced) to 4 (a severe problem).
  The total score thus ranges on a scale between 0-64.
Calcitonin-gene related peptide at baseline (CGRP) | The baseline blood sample was taken up to 7 months after the concussion (4 months median).
  The investigators hypothesized:
  The concentration of calcitonin gene-related peptide (pg/mL) is decreased compared to the healthy control group at baseline
Calcitonin-gene related peptide at follow-up (CGRP) | The follow-up blood sample was taken up to 12 months after baseline (7 months median) after the baseline blood sample.
  The investigators hypothesized:
  The CGRP concentrations (pg/mL) will normalize (increase) at follow-up compared to baseline.

SECONDARY OUTCOMES:
Quinolinic acid at baseline | The baseline blood sample was taken up to 7 months after the concussion (4 months median).
  The investigators hypothesized that:
  The concentration of the neurotoxic metabolite, quinolinic acid (measured in nM), is increased in patients compared to healthy controls
Quinolinic acid at follow-up | The follow-up blood sample was taken up to 12 months after baseline (7 months median) after the baseline blood sample.
  The investigators hypothesized:
  The quinolinic acid concentration (nM) normalizes (decreases) at follow-up compared to the baseline concentration.
Neuroprotective index at baseline | The baseline blood sample was taken up to 7 months after the concussion (4 months median).
  The investigators hypothesized:
  The ratio between the neuroprotective metabolite kynurenic acid (KYNA) and the neurotoxic metabolite quinolinic acid (KynA/QUIN) is lower than the ratio in healthy individuals at baseline.
  A higher ratio means a better outcome.
Neuroprotective index at follow-up | The follow-up blood sample was taken up to 12 months after baseline (7 months median) after the baseline blood sample.
  The investigators hypothesized:
  The ratio between the neuroprotective metabolite kynurenic acid (KYNA) and the neurotoxic metabolite quinolinic acid (QUIN) normalizes (increases) at follow-up compared to baseline. A higher ratio thus means a better outcome.
Inflammatory markers at baseline | The baseline blood sample was taken up to 7 months after the concussion (4 months median).
  The investigators hypothesized that:
  Tumor necrosis factor alpha (TNF-α) and interleukin-6 (IL-6) (both pg/mL) are increased in patients compared to healthy controls.
Inflammatory markers at baseline | The baseline blood sample was taken up to 7 months after the concussion (4 months median).
  The investigators hypothesized:
  Basic fibroblast growth factor (Basic FGF), Eotaxin, interferon gamma (IFN-y), interleukin 1 beta (IL-1B), interleukin 8 (IL-8), interleukin 9 (IL-9), interleukin 17 (IL17), Interferon gamma-induced protein 10 (IP-10), monocyte chemoattractant protein 1 (MCP-1), and Macrophage Inflammatory Protein beta (MIP-1b) (all pg/mL) are significantly increased in patients compared to controls (hypothesis is based on a recent study (PMID: 32326805)
Inflammatory markers at follow-up | The follow-up blood sample was taken up to 12 months after baseline (7 months median) after the baseline blood sample.
  TNF-α and IL-6 (both pg/mL) decreases at follow-up compared to the baseline value in patients.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Preben Eggertsen, MD, Principal Investigator — Hammel Neurorehabilitation Centre and University Research Clinic and Research Unit for Molecular Medicine (Aarhus University)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/42/NCT05812742/SAP_000.pdf